CLINICAL TRIAL: NCT02200822
Title: Systematic Withdrawal of Neurohumoral Blocker Therapy in Optimally Responding Patients to Cardiac Resynchronization Therapy: the STOP-CRT Trial
Brief Title: Systematic Withdrawal of Neurohumoral Blocker Therapy in Optimally Responding CRT Patients
Acronym: STOP-CRT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, MD PhD, MD PhD, Hasselt University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ZOL-STOP-CRT
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure (HF)
Keywords: neurohumoral blocker therapy; renin-angiotensin-aldosterone system (RAAS); RAAS-blocker; beta blocker; spironolactone; angiotensin converting enzyme inhibitor (ACE-I); angiotensin receptor blocker (ARB); cardiac resynchronization therapy (CRT); heart failure; dyssynchrony; left bundle branch block
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-intervention arm (No Intervention): continuation of neurohumoral blocker therapy based on maximum tolerated guideline recommended dose (this group is the control arm for as well withdrawal of beta blocker therapy as withdrawal of RAAS blocker therapy)
- withdrawal of beta blockers (Active Comparator): Intervention arm with systematic withdrawal of beta blocker therapy at a reverse sequence of guideline recommended uptitration.
  (this group is the experimental arm for beta blocker withdrawal. This group receives no intervention with regards to the withdrawal of RAAS blockade). Per 2 weeks:
  * bisoprolol: 10mg/d → 5 mg/d → 2,5 mg/d → 1,25 mg/d stop
  * metoprolol: 200 mg/d → 100 mg/d → 50 mg/d → 25 mg/d → stop
  * nebivolol: 10mg/d → 5 mg/d → 2,5 mg/d → 1,25 mg/d stop
  * carvedilol: 50 mg bid → 25 mg bid → 12,5 mg bid → 6,25 mg bid → stop
  Interventions: Drug: beta blockers
- withdrawal of RAAS blockers (Active Comparator): intervention arm with systematic withdrawal of spironolactone followed by withdrawal of ACE-I/ARB at a reverse sequence of guideline recommended uptitration (this group receives no intervention regarding the withdrawal of beta blockers. This group is the experimental arm for withdrawal of RAAS blockers)
  * first spironolactone/eplerenone: per two weeks: 25 mg/d→12,5 mg/d → stop
  * after 2 weeks stop spironolactone/eplerenone start withdrawal of ACE-I/ARB per two weeks:
    * captopril: 50 mg tid→25 mg tid→12,5 mg tid→6,25 mg tid→stop
    * enalapril: 10 mg bid→5 mg bid→2,5 mg bid→1,25 mg bid→stop
    * lisinopril: 20 mg/d→10 mg/d→5 mg/d→2,5 mg/d→stop
    * ramipril: 10 mg/d→5 mg/d→2,5 mg/d→1,25 mg/d→stop
    * candesartan: 32 mg/d→16 mg/d→8 mg/d→4 m/d→stop
    * valsartan: 160 mg bid→80 mg bid→40 mg bid→20 mg bid→stop
  Interventions: Drug: RAAS blockers
- withdrawal of RAAS - and beta blockers (Active Comparator): intervention arm with systematic withdrawal of spironolactone, secondly ACE-I/ARB and finally beta blockers. (this group is the experimental group for both study interventions (withdrawal of beta blockers and RAAS blockers)
  * First: spironolactone/eplerenone cfr reduction schedule supra
  * After 2 weeks of stop spironolactone withdrawal of ACE-I or ARB cfr reduction schedule supra
  * After 2 weeks of stop ACE-I/ARB withdrawal of beta blocker cfr reduction schedule supra
  Interventions: Drug: beta blockers; Drug: RAAS blockers

INTERVENTIONS:
Drug: beta blockers
  Arms: withdrawal of RAAS - and beta blockers; withdrawal of beta blockers
Drug: RAAS blockers — RAAS blockers (combination of ACE-I/ARB and a mineralocorticoid receptor antagonist)
  Arms: withdrawal of RAAS - and beta blockers; withdrawal of RAAS blockers

SUMMARY:
The primary objective of this study is to demonstrate that in patients with recuperated/normalized left ventricular function, defined as an ejection fraction (EF) ≥ 50%, after implantation of cardiac resynchronization therapy, device treatment is sufficient and neurohumoral blocker therapy can safely be withdrawn

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* CRT implantation

  * based on class I recommendations of ESC (European society of CArdiology) guidelines:
  * Left bundle branch block (LBBB) with QRS duration >150 ms and left ventricular ejection fraction (LVEF) ≤35% who remained NYHA functional class II, III and ambulatory IV despite adequate medical treatment
  * LBBB with QRS duration 120-150 ms and LVEF ≤ 35% who remain in NYHA functional class II, III and ambulatory IV despite adequate medical treatment
* At the moment of inclusion: ≥ 6 months after implantation
* At the moment of inclusion: normalised LVEF (≥ 50%), LVIDD/BSA (left ventricular internal diastolic diameter indexed to body surface area) ≤3.2 cm/m²(woman) en ≤3.1 cm/m² (men) or LVDV/BSA (left ventricular diastolic volume indexed to body surface area) ≤75 ml/m² (women) or ≤75 ml/m² (men)
* euvolemic clinical state and functioning in NYHA class I

Exclusion Criteria:

* contraindication for withdrawal of ACE-I/ARB such as diabetic nephropathy and proteinuria > 1g / 24 h
* severe ventricular arrythmia (sustained VT or ventricular fibrillation) occuring at the time LV function was normalized
* ischemic cardiomyopathy with evidence of scarring (scarring on MRI or severe hypokinesia/akinesia in >1 LV wall segment on echocardiography)
* known severe coronary atherosclerosis (stenosis ≥ 80%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
a > 15% increase in left ventricular end systolic volume | at 12 months

SECONDARY OUTCOMES:
- Incidence of HF related hospitalizations defined as admission to hospital / presentation to emergency room with need for parental therapy | at 12 months
All cause mortality | at 12 months
VO2 max change | at 12 months

OTHER OUTCOMES:
>15% increase in left ventricular end systolic volume | 6 and 24 months
> 15% decrease in left ventricular ejection fraction | at 6, 12 and 24 months
mean blood pressure change | at 6, 12 and 24 months
HF symptoms change (dyspnea visual analogue scale (VAS), New York Heart Association (NYHA) class, questionnaire "Minnesota living with Heart Failure") | at 6, 12 and 24 months
incidence of heart rhythm events (sustained ventricular tachycardia (VT), atrial fibrillation, ventricular fibrillation) | at 6, 12 and 24 months
heart rate variability | at 6, 12 and 24 months
urinary catecholamine concentration | at 6, 12 and 24 months
change in myocardial contractility (force frequence relationship, left ventricular pre-ejection time, iso-volumetric contraction time, dP/dt) | at 6, 12 and 24 months
change in diastolic filling pattern | at 6, 12 and 24 months
plasma concentrations of plasma renin activity and aldosterone | at 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Petra Nijst, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Derived] Nijst P, Martens P, Dauw J, Tang WHW, Bertrand PB, Penders J, Bruckers L, Voros G, Willems R, Vandervoort PM, Dupont M, Mullens W. Withdrawal of Neurohumoral Blockade After Cardiac Resynchronization Therapy. J Am Coll Cardiol. 2020 Mar 31;75(12):1426-1438. doi: 10.1016/j.jacc.2020.01.040. PMID 32216911